CLINICAL TRIAL: NCT05748548
Title: Effects of Lumbal Lordosis and Thoracic Kyphosis Angles on Muscle Activations During Different Low Back Exercises
Brief Title: Effects of Lumbal Lordosis and Thoracic Kyphosis Angles on Muscle Activations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-338
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain, Postural
Keywords: Lumbal Lordosis; Thoracic Kyphosis; Muscle Activations; Low back exercises
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thoracic kyphosis- Lumbal Lordosis angle measurement — In order to determine the kyphosis, the degrees determined by measuring the spinous processes of the T12 T1, T2 and L1 vertebrae with an inclinometer while the individuals are standing will be collected. In order to determine the degree of lumbar lordosis, the measurement between the spinous processes of the T12L1 and S2S3 vertebrae will be made and the degree of lordosis will be determined by adding the degrees found. While the reference values for thoracic kyphosis are 20-45 degrees, this value is 20-40 degrees for lordosis. These measurements will be made with an inclinometer. Measurements will be repeated 3 times and the results will be recorded by taking the average of the measurements.
Other: Back Muscle Endurance Test - Sorenson Test — The endurance of the back muscles will be evaluated with the Biering Sorensen Test (Static Back Endurance Test).
Other: Surface EMG activation — We will try to find out which of the exercises such as pressing back the back, waist extension on the balance ball, lumbar extension while in the active prone position, Superman exercises have better lumbar extensor muscle activations.Muscle activations of individuals will be evaluated using superficial EMG. An 8-channel EMG Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ) will be used to measure signals from the muscles.

SUMMARY:
When the thoracic kyphosis and lumbar lordosis are within a normal range of angular values back pain is less likely to occur. Angular modifications in the physiological curvatures of this sagittal plane have been shown to indicate spinal disorders. For instance, increasing lumbar lordosis and thoracic kyphosis result in higher intradiscal pressure, tension in the spine's passive parts, and creep in the lumbar viscoelastic structures. One of the most important factors of human biomechanics, spinal curvatures provide optimal energy expenditure and movement capacity. Abnormal adaptations in thoracic and lumbar spine biomechanics can cause low back and back pain. Multiple spinal segments are covered by the lumbar erector spinae muscle (LES), which is regarded as a superficial back muscle. LES consists of two muscles, the longissimus thoracis and iliocostalis lumborum. To move the lumbar spine, the lumbar erector spinae muscle (LES) is recruited in a manner that depends on the applied force. It was suggested that patients used LES to compensate for laxity in passive ligamentous structures in an attempt to reduce excessive force on the lumbar spine. Excessive lumbopelvic movements and altered muscle activation patterns are common in patients with low back pain. Researchers have investigated the timing of each muscle's onset and the activity of the LES, and found that patients with low back pain had higher LES activation compared to healthy people. Exercises for strengthening the LES muscle have been performed trunk extension during prone position. Strenghening LES and thoracic extansors may lead to decrease or prevent painful spinal disorders, improve thoracic excessive kyphosis and other complications. Prone trunk extension exercises is used to clinically exercise approcah to activate weak and susceptible to fatigue LES muscle in patients with nonspecific low back pain. This exercise lead to not only strentghening but also lengthening and streching these muscles. To fully understand the effects and underliying the mechanism of this exercise, biomechanical changes in lumbopelvic movement patterns of individuals with kyphotic posture should be examined. Based on current evidence, it is not clear the mechanism that the prone trunk extension exercises is effective on different spinal alignment postures as excessive thoracic khyposis and compansation mechanism on lumbal lordosis. Thus findings from this research may guide clinicians to examine the effects of different prone trunk extension exercises on LES muscles activation. Mitani et al showed that different upper extremity postures effects the lumbal multifudis activations during standing. Brown et al indicated that sit-stand workstations do not change muscle activations of lumbar muscles. Muyor et al concluded that spinal aligment of cyclists affects core muscle activity during cyling. Wattananon et al demonstrated that clinicians should focus on muscle activation patterns rather than the amount of lumbopelvic motion during prone hip extension. Based on the current studies, and to optimally address the underlying mechanism that the main objective was to investigate and show the effects of lumbal lordosis and thoracic kyphosis angles on muscle activations during different low back exercises.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-30
* Individuals who agreed to participate in the study

Exclusion Criteria:

* Individuals with congenital lumbar pathology
* Individuals who have previously had an operation on the back and waist region
* Individuals with scoliosis
* Individuals with a difference in length in the lower extremity

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Individuals who agreed to participate in the study were determined as individuals between the ages of 18-30.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-22 (Estimated); Primary Completion 2023-04-22 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Surface EMG activation | 4 weeks
  The investigators will try to find out which of the exercises such as pressing the back back, waist extension on the balance ball, lumbar extension in the active prone position, Superman exercises have better lumbar extensor muscle activations. Muscle activations of individuals will be evaluated using superficial EMG. An 8-channel EMG Noraxon MiniDTS system (Noraxon, USA, Inc., Scottsdale, AZ) will be used to measure signals from the muscles.
Thoracic kyphosis- Lumbal Lordosis angle measurement | 4 weeks
  In order to determine the kyphosis, the degrees determined by measuring the spinous processes of the T12 T1, T2 and L1 vertebrae with an inclinometer while the individuals are standing will be collected. In order to determine the degree of lumbar lordosis, the measurement between the spinous processes of the T12L1 and S2S3 vertebrae will be made and the degree of lordosis will be determined by adding the degrees found. While the reference values for thoracic kyphosis are 20-45 degrees, this value is 20-40 degrees for lordosis. These measurements will be made with an inclinometer. Measurements will be repeated 3 times and the results will be recorded by taking the average of the measurements.
Back Muscle Endurance Test - Sorenson Test | 4 weeks
  The endurance of the back muscles will be evaluated with the Biering Sorensen Test (Static Back Endurance Test).

CONTACTS AND LOCATIONS:
Overall Officials: Caglar Soylu, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided